CLINICAL TRIAL: NCT02526667
Title: Assessment of the Antimicrobial Efficacy of 2% CHG Cloth Preoperative Skin Preparation
Brief Title: Preoperative Chlorhexidine Gluconate (CHG) Cloth on Healthy Volunteers
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Medline Industries (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: R15-029
Record Dates: First submitted 2015-08-16; First posted 2015-08-18 (Estimated); Results first posted 2020-09-28 (Actual); Last update posted 2020-09-28 (Actual); Status verified 2020-09

CONDITIONS: Surgery
Keywords: Preoperative surgical skin preparation
MeSH Terms: interventions — chlorhexidine gluconate

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Chlorhexidine Gluconate Cloth (Experimental): 2% CHG, single application
  Interventions: Drug: Chlorhexidine gluconate
- Vehicle Cloth (Placebo Comparator): Excipients on cloth
  Interventions: Other: Vehicle
- Active Chlorhexidine gluconate solution (Active Comparator): Dynahex 2% CHG
  Interventions: Drug: DynaHex-2

INTERVENTIONS:
Drug: Chlorhexidine gluconate — 2% CHG solution on cloth
  Other Names: CHG
  Arms: Chlorhexidine Gluconate Cloth
Drug: DynaHex-2 — 2% CHG solution
  Other Names: CHG 2%
  Arms: Active Chlorhexidine gluconate solution
Other: Vehicle — Excipients of CHG product only
  Other Names: Control
  Arms: Vehicle Cloth

SUMMARY:
Evaluate the effects of Chlorhexidine Gluconate (CHG) cloth on the reduction of bacteria on the skin.

DETAILED DESCRIPTION:
Examine the antimicrobial cloth effects on normal flora bacteria of the abdomen and groin areas post Chlorhexidine Gluconate (CHG) application.

ELIGIBILITY:
Inclusion Criteria:

* Males or Females
* 18 years of age or older
* Signed informed consent
* Good Health
* Six inches of abdomen and groin areas without tattoos, or skin disorders

Exclusion Criteria:

* Dermatological Conditions
* Sensitivity to latex
* Sensitivity to CHG

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 340 (Actual)
Dates: Start 2015-08; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: R Olsavcszky, MD, Principal Investigator — S.C. BIO HIGH TECH S.R.L.
Locations (1):
- Bio High Tech SRL, Bucharest, Romania

IPD SHARING:
Plan to Share IPD: Yes
Data to be shared with FDA.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Upon achieving sufficient microbial growth prior to product application on either the abdomen, groin or both abdomen and groin regions,sites of the participant were then randomized to receive one or two products for evaluation for up to 4 sites. Differences in the number of participants is based on microbial qualification.
Pre-assignment Details: The sites of the participant were tested for microbial activity after product application. In some instances, more than one product could have been applied to a participant but only one product per site (groin and/or abdomen sites). Up to 4 sites could be treated: 1) both groin and abdomen, 2) only the groin or 3) only the abdomen.
Units Other Than Participants: Sites
Groups:
- CHG Cloth: CHG, 3 min application
- Vehicle: Vehicle 3 min application
- Comparator CHG: CHG comparator application
Period: Abdomen
Arm/Group | CHG Cloth | Vehicle | Comparator CHG
Started | 284; 568 Sites | 56; 112 Sites | 281; 562 Sites
Completed | 284; 307 Sites | 56; 59 Sites | 281; 314 Sites
Not Completed | 0; 261 Sites | 0; 53 Sites | 0; 248 Sites
Period: Groin
Arm/Group | CHG Cloth | Vehicle | Comparator CHG
Started | 290; 580 Sites | 56; 112 Sites | 294; 588 Sites
Completed | 290; 291 Sites | 56; 55 Sites | 294; 294 Sites
Not Completed | 0; 289 Sites | 0; 57 Sites | 0; 294 Sites

BASELINE CHARACTERISTICS:
Groups:
- CHG, Vehicle, Comparator CHG: Single applications of products. 3 min application for CHG and Vehicle. Comparator CHG applied according to instructions.
Arm/Group | CHG, Vehicle, Comparator CHG
Number analyzed (Participants) | 340
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1
  Between 18 and 65 years | 315
  >=65 years | 24
Age, Continuous [Mean (Full Range); unit: years] | 38 [18 to 69]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 182
  Male | 158
Region of Enrollment [Number; unit: participants]
  Romania | 340

OUTCOME MEASURES:

1. Primary Outcome: Responder Rates (%) of Sites Identified for Bacterial Reduction on the Abdomen and Groin
Description: Log10 reduction in bacteria on the skin evaluated at 10 minutes, 6 hours and 8 hours after treatment. Responder rates (%) are the percentage of sites identified that produced a 2-Log and 3-Log reduction from baseline for abdomen and groin sites respectively.
Time Frame: 10 minutes, 6 hours, 8 hours
Population: Number of participants involved in the analyses.
Measure: Number; unit: Percent of sites
Units Other Than Participants: Sites
Groups:
- CHG 3 Min Abdomen; Vehicle Abdomen; Comparator CHG Abdomen: single application on abdomen
- CHG 3 Min Groin; Vehicle Groin; Comparator CHG Groin: single application on groin
Arm/Group | CHG 3 Min Abdomen | CHG 3 Min Groin | Vehicle Abdomen | Vehicle Groin | Comparator CHG Abdomen | Comparator CHG Groin
Number analyzed (Participants) | 284 | 290 | 56 | 56 | 281 | 294
Number analyzed (Sites) | 307 | 291 | 59 | 55 | 314 | 294
Percent of sites
  10 min | 78 | 84 | 54 | 56 | 72 | 73
  6 hours | 100 | 100 | 96 | 100 | 99 | 100
  8 hours | 99 | 100 | 96 | 100 | 98 | 100

ADVERSE EVENTS:
Groups:
- CHG Cloth Abdomen: CHG, 3 min application to abdomen
- Vehicle Abdomen: Vehicle 3 min application to abdomen
- Comparator CHG Abdomen: CHG comparator applied to abdomen
- CHG Cloth Groin: CHG, 3 min application to groin
- Vehicle Groin: Vehicle 3 min application to groin
- Comparator CHG Groin: CHG comparator applied to groin
Arm/Group | CHG Cloth Abdomen | Vehicle Abdomen | Comparator CHG Abdomen | CHG Cloth Groin | Vehicle Groin | Comparator CHG Groin
Serious Adverse Events (participants affected / at risk) | 0/284 | 0/56 | 0/281 | 0/290 | 0/56 | 0/294
Other Adverse Events (participants affected / at risk) | 0/284 | 0/56 | 0/281 | 0/290 | 0/56 | 0/294

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Confidential information based on contract.